CLINICAL TRIAL: NCT06066879
Title: Non Randomized Cohort Study to Evaluate Pre-operative Ketamine Infusion for the Decrease Overall Pain Levels Following Revision Cervical or Lumbar Fusion Surgery Through the Post-operative Phase, Decreasing Reliance on Opioids for Daily Pain Control, Opioid Related Adverse Events, as Well as Improving Mood, Functionality, and Quality of Life for Patients That Live With Chronic Pain Syndromes.
Brief Title: Pre-Operative Ketamine Infusion for Post Operative Pain Control After Revision Spinal Surgery
Acronym: KIPSs
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AXIS Spine Center- a division of Northwest Specialty Hospital (Other)
Collaborators: IDAHO PANHANDLE HEALTH DISTRICT (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPS001
Record Dates: First submitted 2023-09-28; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Revision Spine Surgery; Fusion of Spine; Cervical Fusion; Lumbar Fusion
Keywords: ketamine; revision surgery; opioid
MeSH Terms: conditions — Klippel-Feil Syndrome | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Infusion (Experimental): ketamine infusion at 0.5 mg/kg over one hour two weeks (14 days) prior to their scheduled surgical date
  Interventions: Drug: Ketamine Hydrochloride
- Standard Of Care (No Intervention): No use of ketamine pre, intra, or post-operatively

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Pre-Operative Ketamine infusion
  Arms: Ketamine Infusion

SUMMARY:
To determine if a pre-operative ketamine infusion would provide a similar decrease in post-operative analgesic and opioid consumption as intra-operative ketamine, but expand the monitoring period through the post-operative phase up to 90 days. Hypothesis is that pre-operative ketamine infusion will lead to a decrease in narcotic consumption from baseline following an elective cervical or lumbar fusion, leading to increased functionality and quality of life for these patients.

DETAILED DESCRIPTION:
Patients with chronic pain requiring daily opioid use for pain control turn to invasive surgeries for long-term management of their pain, though there is still a chance of requiring opioid pain medications as well as increased use during the immediate post-operative phase. Ketamine infusion peri-operatively has been shown to decrease post-operative pain from invasive surgeries, such as cervical and lumbar fusions, and there is also evidence that ketamine infusions in general can help to improve levels of chronic pain with less need for opioid medications. Our study asks if pre-operative ketamine infusion will decrease overall pain levels following cervical or lumbar surgery through the post-operative phase, decreasing reliance on opioids for daily pain control, as well as improving mood, functionality, and quality of life for patients that live with chronic pain syndromes. Ketamine, an N-methyl-D-aspartate receptor antagonist, has newly received attention for its ability to provide anesthesia in patients with chronic pain syndromes and neuropathic pain syndromes. Recent studies have shown evidence that intra-operative delivery of ketamine can reduce acute post-operative analgesic consumption in patients following a variety of surgical procedures, though this is often focused on the acute post-operative period (initial 72 hours). Additionally, studies have shown that ketamine infusions in patients with chronic pain requiring opioid analgesics does provide some variable level of baseline pain improvement. For patients with chronic neck or back pain, choosing to undergo invasive spinal surgeries potentially could provide some relief of their daily pain, though there is a chance that they will still require daily narcotics for pain relief post-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18-75
2. Able to understand the informed consent form and provide written informed consent and able to complete outcome measures
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Daily opiate use totaling ≥50 morphine milli-equivalents (MME) or more for 6 weeks or greater
5. Scheduled for revision surgical fusion of the cervical or lumbar spine
6. Total duration of neck or back pain >12 weeks

Exclusion Criteria:

1. Current use of Ketamine for any other medical conditions
2. Uncontrolled hypertension
3. Uncontrolled Diabetes
4. Increased intracranial pressure
5. Pregnancy or lactation
6. Known allergic reactions to components of ketamine or midazolam
7. Participants who ultimately require intra-operative ketamine administration for anesthesia
8. Treatment with another investigational drug or other intervention within 12 months of study treatment
9. History of psychosis or schizophrenia
10. History of conversion disorder
11. History of clotting disease
12. Pending or active compensation claim, litigation or disability remuneration (secondary gain)
13. Surgically naïve patients
14. Allergies to any of the medications to be used during the procedures
15. Active infection or systemic or localized infection at needle entry sites (subject may be considered for inclusion once infection is resolved)
16. Uncontrolled immunosuppression (e.g. AIDS, cancer)
17. Participating in another clinical trial/investigation within 30 days prior to signing informed consent
18. Subject unwilling or unable to comply with follow up schedule or protocol requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Degree of reduction in opiate consumption following surgery | 12 weeks

SECONDARY OUTCOMES:
Responder rate | 12 weeks
  The proportion of subjects who experience at least 50% reduction in back pain intensity (improvement in ODI scores) at 3 months as compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Jameson, MD, Principal Investigator — division of NSWH
Locations (1):
- AXIS Spine, Coeur d'Alene, Idaho, United States

IPD SHARING:
Plan to Share IPD: Undecided